CLINICAL TRIAL: NCT03315494
Title: A Phase 1, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Multiple Oral Doses of SKI-O-703 in Healthy Volunteers
Brief Title: Safety, Tolerability, and Pharmacokinetics of Multiple Ascending Doses of SKI-O-703 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oscotec Inc. (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSCO-P1202
Record Dates: First submitted 2017-10-06; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: Arthritis, Rheumatoid
Keywords: rheumatoid arthritis; healthy volunteers; moderate to severe
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — cevidoplenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- SKI-O-703 200 mg (once daily) (Experimental): SKI-O-703 capsule (1 x 200 mg)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 400 mg (once daily) (Experimental): SKI-O-703 capsule (2 x 200 mg, once daily)
  Interventions: Drug: SKI-O-703 capsule
- SKI-O-703 200 mg (twice daily) (Experimental): SKI-O-703 capsule (1 x 200 mg twice daily)
  Interventions: Drug: SKI-O-703 capsule
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo capsule

INTERVENTIONS:
Drug: SKI-O-703 capsule — SKI-O-703 200 mg capsule with no inactive excipients.
  Arms: SKI-O-703 200 mg (once daily); SKI-O-703 200 mg (twice daily); SKI-O-703 400 mg (once daily)
Drug: Placebo capsule — Placebo 180 mg capsule filled with microcrystalline cellulose.
  Arms: Placebo

SUMMARY:
This double-blind, placebo-controlled, multiple ascending dose study is designed to evaluate the safety, tolerability, and pharmacokinetics (PK) of SKI-O-703 in healthy volunteers.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled study in healthy adult volunteers, to evaluate the safety, tolerability, and pharmacokinetics (PK) of multiple ascending doses of SKI-O-703. A total of 24 subjects are planned to participate in 3 cohorts (8 subjects each). In each cohort, 6 subjects will be randomly assigned to receive SKI-O-703 and 2 subjects will be randomly assigned to matching placebo. Dosing will be initiated with a 200 mg once daily (QD) dose cohort and escalated to 400 mg QD, under fasting conditions, for 7 days. In the third cohort, a 200 mg twice daily (BID) dose will be studied for 7 days. Evening dosing will occur 12 hours after the morning dose and will be preceded by fasting for at least 3 hours. After all 8 subjects in each cohort have received the study drug and been monitored, the decision to escalate to the next dose cohort will be made.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for participation prior to completing any study procedures.
* Considered by investigator to be in good health, as judged by absence of clinically significant diseases and clinically significant abnormal values as determined by detailed medical history review, complete physical examination, and clinical laboratory evaluations.
* Male subjects and female subjects of non-childbearing potential 18-55 years old, inclusive, at time of screening.
* Females of non-childbearing potential are those who have been surgically sterile for at least 6 months or who have been postmenopausal for at least 2 years and have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
* Male subjects agree to use a condom with spermicide or to abstain from sexual intercourse for 90 days after dosing.
* Male subjects must agree not to donate sperm for 90 days after dosing.
* Female subjects must have negative pregnancy tests at screening and on Day -1.
* Body mass index between 18.0 and 30.0 kg/m2, inclusive, and body weight of ≥ 50 kg.
* Able to understand the study and any risks of participation and able to communicate with the investigator.

Exclusion Criteria:

* History of any clinically significant disease or disorder that may put the subject at risk due to study participation, impact the subject's ability to participate in the study, or influence the study results.
* History or presence of any gastrointestinal, hepatic or renal disease or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
* Any surgical or medical condition that could possibly affect drug absorption, distribution, metabolism, and excretion (e.g. bariatric procedure).
* Any medical/surgical procedure or trauma within 4 weeks prior to Day -1 as determined by the investigator.
* Any clinically significant infection within 3 months prior to Day -1 as determined by the investigator.
* Any of the following abnormal laboratory values upon repeat testing at Screening or Check-in (Day -1):

  1. Hemoglobin < lower limit of normal (LLN),
  2. Platelet count <LLN,
  3. Absolute neutrophil count <LLN or >upper limit of normal (ULN),
  4. Alanine aminotransferase or aspartate aminotransferase >ULN,
  5. Creatinine or blood urea nitrogen >ULN, or
  6. Any other clinically significant, in the opinion of the investigator, abnormal laboratory result.
* Use of concomitant medications from 30 days or 5 half-lives prior to Day -1 (whichever is longer) through completion of the End of Study (EOS) visit, including prescription medications, nutritional supplements, herbal remedies, and over-the-counter medications (note: use of vitamin supplements should be stopped at least 7 days prior to Screening through completion of the EOS visit).
* Receipt of any investigational medication within 30 days or 5 half-lives prior to Day -1, whichever is longer.
* Use of tobacco or nicotine-containing products within 30 days prior to Day -1 through the EOS visit.
* Use of CYP3A inducers and inhibitors (including St. John's wort) within 30 days prior to dosing.
* Intake of food or beverage containing alcohol, grapefruit or grapefruit juice, apple or orange juice, vegetables from the mustard green family (e.g. kale, broccoli, watercress, collard greens, kohlrabi, Brussels sprouts, mustard), or charbroiled meats within 1 week prior to dosing.
* History of substance abuse, drug addiction, or alcoholism.
* Positive urine drug or urine alcohol test at Screening or Day -1 or unable to abstain from alcohol from 72 hours prior to study entry through the EOS visit.
* Unable to abstain from caffeine- and xanthine-containing products from 72 hours prior to dosing through discharge from the study center.
* Female subjects who are pregnant or lactating or have a positive pregnancy test at Screening or Day -1.
* Positive result at Screening for human immunodeficiency virus, hepatitis B surface antigen, or hepatitis C virus antibody or positive result for hepatitis B core antibody with a negative result for hepatitis B surface antigen.
* Recent (within the past 5 years) history of malignancy, except successfully treated basal cell carcinoma.
* High blood pressure, defined as >140 mm Hg systolic blood pressure or >90 mm Hg diastolic blood pressure upon repeat confirmation (repeated up to 4 times).
* Cardiac arrhythmias or clinically significant electrocardiogram (ECG) findings.
* Corrected QT interval >450 milliseconds or deemed clinically significant by the investigator (may be repeated for confirmation).
* Family history of long QT syndrome.
* Blood loss or blood donation >450 mL within 4 weeks prior to study drug dosing.
* History of sensitivity to drugs with chemical similarity to the study medication, its components, or the excipients.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-09-22 (Actual); Primary Completion 2016-12-21 (Actual); Study Completion 2016-12-21 (Actual)

PRIMARY OUTCOMES:
Number of participants (Healthy Volunteers) with reported adverse events receiving multiple dose of SKI-O-703 as assessment of safety and tolerability. | 21 days
  Safety and tolerability of SKI-O-703 as measured by subject incidence of treatment-related Adverse Events.

SECONDARY OUTCOMES:
Area under the concentration versus time curve within a dosing interval (AUC0-tau), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  AUC0-tau will be reported.
Area under the concentration versus time curve from time 0 to the last measurable concentration (AUC0-t), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  AUC0-t will be reported.
Area under the concentration versus time curve within a dosing interval (AUC0-inf), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Day 7 only
  AUC0-inf will be reported.
Maximum observed concentration (Cmax), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  Cmax will be reported.
Apparent oral clearance (CL/F), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  CL/F will be reported.
Terminal elimination rate constant (Kel), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Day 7
  Kel will be reported.
Time to reach the maximum observed concentration, to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  Tmax will be reported.
Apparent terminal elimination half-life (t1/2), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Day 7 only
  t1/2 will be reported.
Apparent volume of distribution (Vd/F), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  Vd/F will be reported.
Metabolite ratio (Rmet), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  Rmet will be reported.
Accumulation ratio based on AUC0-tau (RAUC), to investigate pharmacokinetic profiles of SKI-O-592 (the free base of SKI-O-703) and its metabolites (M2 and M4) in healthy volunteers. | Days 1-7 (dosing), post-dose (days 8-10).
  RAUC will be reported.

OTHER OUTCOMES:
The pharmacodynamics variable will be the change in the percentage of activated gp53/CD63+ basophils and will be evaluated from serial blood samples collected from subjects who have received SKI-O-703 or placebo. | Days 1-7 (dosing), post-dose (day 8).
  Changes in the percentage of activated gp53/CD63+ basophils will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- PPD Development, LP, Austin, Texas, United States